CLINICAL TRIAL: NCT02033356
Title: An Estimate of the ED95 of Lidocaine 1.0% for Filling the Adductor Canal When Placing an Adductor Canal Block in Healthy Volunteers
Brief Title: ED95 of Lidocaine 1.0% for Filling the Adductor Canal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Pia Jaeger, MD, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM3-PJ-13; 2013-004462-33 (EudraCT Number)
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: adductor canal block; volunteers; US-guided peripheral nerve block; lower limb; MRI
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- ACB with 30 ml lidocaine 1% (Experimental): Procedure/Surgery: Adductor canal block with lidocaine 1% The Continual Reassessment Method is used to calculate the dose level consecutively for every new cohort (2 subjects) in the study.
  Possible dose levels are: 5, 10, 15, 20, 25 and 30 ml.
  Interventions: Procedure: Adductor canal block with lidocaine 1%; Drug: Lidocaine
- ACB with 25 ml lidocaine 1% (Experimental): Procedure/Surgery: Adductor canal block with lidocaine 1% The Continual Reassessment Method is used to calculate the dose level consecutively for every new cohort (2 subjects) in the study.
  Possible dose levels are: 5, 10, 15, 20, 25 and 30 ml.
  Interventions: Procedure: Adductor canal block with lidocaine 1%; Drug: Lidocaine
- ACB with 20 ml lidocaine 1% (Experimental): Procedure/Surgery: Adductor canal block with lidocaine 1% The Continual Reassessment Method is used to calculate the dose level consecutively for every new cohort (2 subjects) in the study.
  Possible dose levels are: 5, 10, 15, 20, 25 and 30 ml.
  Interventions: Procedure: Adductor canal block with lidocaine 1%; Drug: Lidocaine
- ACB with 15 ml lidocaine 1% (Experimental): Procedure/Surgery: Adductor canal block with lidocaine 1% The Continual Reassessment Method is used to calculate the dose level consecutively for every new cohort (2 subjects) in the study.
  Possible dose levels are: 5, 10, 15, 20, 25 and 30 ml.
  Interventions: Procedure: Adductor canal block with lidocaine 1%; Drug: Lidocaine
- ACB with 10 ml lidocaine 1% (Experimental): Procedure/Surgery: Adductor canal block with lidocaine 1% The Continual Reassessment Method is used to calculate the dose level consecutively for every new cohort (2 subjects) in the study.
  Possible dose levels are: 5, 10, 15, 20, 25 and 30 ml.
  Interventions: Procedure: Adductor canal block with lidocaine 1%; Drug: Lidocaine
- ACB with 5 ml lidocaine 1% (Experimental): Procedure/Surgery: Adductor canal block with lidocaine 1% The Continual Reassessment Method is used to calculate the dose level consecutively for every new cohort (2 subjects) in the study.
  Possible dose levels are: 5, 10, 15, 20, 25 and 30 ml.
  Interventions: Procedure: Adductor canal block with lidocaine 1%; Drug: Lidocaine

INTERVENTIONS:
Procedure: Adductor canal block with lidocaine 1% — US-guided adductor canal block
Drug: Lidocaine

SUMMARY:
The aim of this prospective dose finding study is to estimate the minimal effective volume (ED95) for lidocaine 1.0% for filling the adductor canal when placing an adductor canal block. We will apply the Continual Reassessment Method (CRM) for estimating the ED95 and use an MRI scan to evaluate the main objective and ensure spread to the distal part of the adductor canal.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years
* Men
* American Society of Anesthesiologists' class 1
* Body Mass Index 18-25

Exclusion Criteria:

* Allergy to study medication
* Earlier trauma or surgery to the lower limb
* Diabetes Mellitus - Contraindications to MRI

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To estimate the ED 95 for the volume needed to fill the adductor canal distally. | MRI performed 15 minutes post block
  This will be evaluated as a binary outcome using MRI; where the adductor canal is considered to be filled if the lidocaine injectate can be identified inside the canal in the first slice distally to the insertion of the adductor longus muscle on femur.

SECONDARY OUTCOMES:
To investigate the effect of volume on proximal spread to the femoral triangle | MRI performed 15 minutes post block
  Evaluated as a binary outcome using MRI
Quadriceps muscle strength | 1 hour post block
  To investigate the effect of volume on quadriceps muscle strength, assessed as maximum voluntary isometric contraction (MVIC) and evaluated as a binary outcome (reduction by more or less than 25%).
Pin prick test | 1 hour post block
  To investigate the effect of volume on sensory block assessed by pin-prick in the saphenous innervation area and in the popliteal fossa.
Temperature discrimination test | 1 hour post block
  To investigate the effect of volume on sensory block assessed by cold sensation using alchohol swabs, in the saphenous innervation area and in the popliteal fossa.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jaeger, MD, Principal Investigator — Department of Anaesthesia, HOC, Rigshospitalet, Denmark
Locations (1):
- Aleris-Hamlet Hospitals Copenhagen, Søborg, Denmark

REFERENCES:
- [Derived] Jaeger P, Jenstrup MT, Lund J, Siersma V, Brondum V, Hilsted KL, Dahl JB. Optimal volume of local anaesthetic for adductor canal block: using the continual reassessment method to estimate ED95. Br J Anaesth. 2015 Dec;115(6):920-6. doi: 10.1093/bja/aev362. PMID 26582853